CLINICAL TRIAL: NCT00437385
Title: Phase 1 Study: Evaluation of Three Continuation Therapies After Acute Electroconvusive Therapy (ECT) Concerning Efficacy and Cognition in Severly Depressed Patients
Brief Title: Evaluation of Three Continuation Therapies After ECT Concerning Efficacy and Cognition in Severly Depressed Patients
Acronym: EffECT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Eva-Lotta Brakemeier, Dr. rer. nat., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ek224-05b
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Depression; Major Depression
Keywords: therapy resistant depression, severe depression
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Selective Serotonin Reuptake Inhibitors; Serotonin and Noradrenaline Reuptake Inhibitors; Lithium; Electroconvulsive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Continuation-Medication with Antidepressants (after WBS Guidelines)
  Interventions: Drug: TCAs, SSRIs, NARIs, SNRIs, Lithium
- 2 (Experimental): Continuation-ECT with Antidepressants
  Interventions: Drug: TCAs, SSRIs, NARIs, SNRIs, Lithium; Procedure: Electroconvulsive therapy
- 3 (Experimental): Continuation-Psychotherapy (Cognitive Behavioral Group Psychotherapy including the "Situational Analysis" of CBASP)
  Interventions: Drug: TCAs, SSRIs, NARIs, SNRIs, Lithium; Behavioral: Cognitive behavioral group therapy

INTERVENTIONS:
Drug: TCAs, SSRIs, NARIs, SNRIs, Lithium — Antidepressant, dosage, and duration are chosen due to the guidelines of the WFSBP (Bauer et al. 2002)
Procedure: Electroconvulsive therapy — ECT treatment is administered three times per week on non-successive weekdays and according to existing standards. Treatment lasts for at least three weeks (nine ECT sessions). Psychopharmacological treatment is continued during ECT treatment. Patients receive ultrabrief pulse (0.3 ms), unilateral treatment at a frequency of 40-100 Hertz. Stimulation is applied to the non-dominant hemisphere, according to the d'Elia electrode positioning paradigm. All patients are initially treated with right unilateral stimulation and in case of non-response switched to bilateral treatment. Stimulus intensity is chosen according to individual seizure threshold and administered at 2.5 to 6-fold intensity. During the ECT session, patients are anesthetized, under the influence of a muscle relaxant, and monitored regarding their vital functions.
  Arms: 2
Behavioral: Cognitive behavioral group therapy — The continuation-psychotherapy (continuation cognitive behavioral therapy, C-CBT) sample took part in a newly developed cognitive behavioral group therapy program called "EffECTive". This therapy program was developed within the EffECT-project (Brakemeier et al. 2005), to fit the specific target group of patients finished with acute ECT-treatment. EffECTive is a group therapy that combines several aspects of existing cognitive-behavioral depression manuals with new elements (e.g., the situational analysis from CBASP, McCullough 2000), to fit the target group. Therapy sessions were held once a week and include approximately 15 sessions until follow-up.
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate three different continuation treatments after acute ECT concerning efficacy and impact on cognition in severly depressed patients.

DETAILED DESCRIPTION:
BACKGROUND While electroconvulsive therapy (ECT) in major depression is effective, high relapse rates and cognitive effects limit its long-term use. Continuation treatment after ECT with combinations of C-ECT or psychotherapy and medication may decrease relapse rates and cognitive side effects while changing cognitive psychological variables like dysfunctional attitudes in the long-term.

CENTRAL RESEARCH QUESTIONS

* Evaluation of the efficacy of three continuation treatments aimed at preventing relapses after acute ECT
* Examination of the cognitive side effects and the changes of cognitive psychological variables during acute and continuation treatment

METHODS In a prospective, randomized, controlled, long-term study we assign 60 depressed ECT responder either to antidepressant treatment alone, or C-ECT plus medication, or cognitive behavioral group therapy plus medication. Depressive symptoms and cognition were assessed before, during, immediately after acute ECT and two, four, six, and 12 months during continuation therapy.

HYPOTHESES It is hypothesized that the use of combination continuation therapies after effective ECT leads to lower HAMD scores and lower relapse rates than the standard treatment with antidepressants alone after 6 months. In addition, we assume that the CBT group will establish more functional macro-patterns than the somatic treatments in the long term and will have the lowest HAMD scores and relapse rates after 1 year. With regard to the cognitive side effects, the autobiographical memory is expected to be the only specific part of memory being affected negatively by ECT in the short and long term.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive episode (unipolar)
* Response to acute ECT (at least 50% reduction in HAMD)
* Capacity to consent
* Sufficient comprehension of the German language

Exclusion Criteria:

* Schizophrenia, schizoaffective disorder, or other psychosis
* Amnestic disorder, dementia, or delirium
* Pregnancy
* Epilepsy
* Current alcohol or substance abuse or dependence
* CNS disease or brain injury not associated with psychotropic drug exposure
* ECT in the past 3 months
* Acute suicidality
* Judiciary hospitalization

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2005-03; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Score on HAMD after 6 and 12 months | 6 and 12 months after enetering continuation phase

SECONDARY OUTCOMES:
Relapse rate after 6 and 12 months | 6 and 12 months after enetering continuation phase
Response and remission rates after 6 and 12 months | 6 and 12 months after enetering continuation phase
Scores on MADRS, BDI, and CGI after 6 and 12 months | 6 and 12 months after enetering continuation phase

CONTACTS AND LOCATIONS:
Overall Officials: Malek Bajbouj, PhD, Study Chair — Department of Psychiatry, Charité University Medicine, Campus Benjamin Franklin, Berlin, Germany; Eva-Lotta Brakemeier, MA, Principal Investigator — Department of Psychiatry and Psychotherapy, University Medicine, Freiburg, Germany; Norbert Kathmann, PhD, Study Chair — Department of Clinical Psychology, Humboldt-University, Berlin, Germany
Locations (1):
- Department of Psychiatry, Charité University Medicine, Campus Benjamin Franklin, Berlin, Germany, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Sackeim HA, Haskett RF, Mulsant BH, Thase ME, Mann JJ, Pettinati HM, Greenberg RM, Crowe RR, Cooper TB, Prudic J. Continuation pharmacotherapy in the prevention of relapse following electroconvulsive therapy: a randomized controlled trial. JAMA. 2001 Mar 14;285(10):1299-307. doi: 10.1001/jama.285.10.1299. PMID 11255384
- [Background] Lisanby SH, Maddox JH, Prudic J, Devanand DP, Sackeim HA. The effects of electroconvulsive therapy on memory of autobiographical and public events. Arch Gen Psychiatry. 2000 Jun;57(6):581-90. doi: 10.1001/archpsyc.57.6.581. PMID 10839336
- [Background] Kellner CH, Knapp RG, Petrides G, Rummans TA, Husain MM, Rasmussen K, Mueller M, Bernstein HJ, O'Connor K, Smith G, Biggs M, Bailine SH, Malur C, Yim E, McClintock S, Sampson S, Fink M. Continuation electroconvulsive therapy vs pharmacotherapy for relapse prevention in major depression: a multisite study from the Consortium for Research in Electroconvulsive Therapy (CORE). Arch Gen Psychiatry. 2006 Dec;63(12):1337-44. doi: 10.1001/archpsyc.63.12.1337. PMID 17146008
- [Derived] Brakemeier EL, Merkl A, Wilbertz G, Quante A, Regen F, Buhrsch N, van Hall F, Kischkel E, Danker-Hopfe H, Anghelescu I, Heuser I, Kathmann N, Bajbouj M. Cognitive-behavioral therapy as continuation treatment to sustain response after electroconvulsive therapy in depression: a randomized controlled trial. Biol Psychiatry. 2014 Aug 1;76(3):194-202. doi: 10.1016/j.biopsych.2013.11.030. Epub 2013 Dec 12. PMID 24462229
- See also: Related Info — http://www.charite-psychiatrie.de/menue-links/module/affektive-stoerungen/as-forschungsschwerp.html